CLINICAL TRIAL: NCT04021251
Title: Performance Characteristics of Non-invasive Glucose Monitoring Device Prototypes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-16
Record Dates: First submitted 2018-12-20; First posted 2019-07-16 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Short term collection of IMD data (Experimental): Subjects will collect spectral raman data on P0.2 for minimum 10 hours per day with a maximum of 15 minutes between each measurement for 5 days distributed over a time period of 10 days. Spectral data will be compared to standard BG and/or FGM measurements.
  Interventions: Device: P0.2
- Medium term collection of IMD data (Experimental): Subjects will collect spectral raman data on P0.2 for four times a day for 30 days distributed over a time period of 40 days. Spectral data will be compared to standard BG measurements.
  Interventions: Device: P0.2
- Long term collection of IMD data (Experimental): Subjects will collect spectral raman data on P0.2 for four times a day for 90 days distributed over a time period of 6 months. Spectral data will be compared to standard BG measurements.
  Interventions: Device: P0.2
- Medium term collection of IMD data, increased # of sessions (Experimental): Subjects will collect spectral raman data on P0.2 four times a day for 30 days distributed over a time period of 40 days. Spectral data will be compared to standard BG measurements. The number of optical sessions performed each time measurements are done are increased compared to the investigation's second arm.
  Interventions: Device: P0.2

INTERVENTIONS:
Device: P0.2 — Investigational Medical Device collecting spectral raman data from tissue.

SUMMARY:
This clinical study has been launched to collect spectral raman data paired with validated glucose reference values in private homes of subjects

DETAILED DESCRIPTION:
Subjects will collect either 8 or 44 daily optical raman readings paired with either 8 capillary Blood Glucose comparator or 8 capillary Blood Glucose comparator plus 44 readings using a flash glucose monitoring system in own home with maintaining usual routines. Subjects will either collect data for 5 days during a 10 days period or collect data for 90 days during a 40 days period or collect data for 90 days during 6 months period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older
* Diabetic patients (all types)
* Skin phototype 1-4

Exclusion Criteria:

* For female participants: Pregnancy or subject is attempting to conceive or not willing and able to practice birth control during the study duration
* For female participants: Breastfeeding
* Subjects not able to understand and read Danish
* In Investigator's opinion, subject is not able to follow instructions as specified in the protocol
* Participants not able to hold hand/arm steadily (including tremors and Parkinson's Disease)
* Diagnosed with reduced circulation
* Extensive skin changes, tattoos or diseases on probe application site
* Known allergy to medical grade alcohol
* Known allergy to adhesives, applicable to subjects in RSP-16-01
* Systemic or topical administration of glucocorticoids for the past 7 days and under investigation
* Participants undergoing dialysis treatment
* Medical history or any condition that may, in the opinion of the Investigator, compromise the subject's ability to participate
* Concomitant medical condition which could present a risk to the safety or welfare of the subject or study staff.
* Participants currently enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Generation of predictive algorithms for determining blood glucose levels | 3 years
  Collected spectral raman data will found the development of predictive algorithms for glucose determination.
Validation of predictive algorithms for determining blood glucose levels | 3 years
  Performance of predictive models will be evaluated using the consensus error grid.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Erik Henriksen, MD, Principal Investigator — Odense University Hospital, Dpt. of Endocrinology M
Locations (1):
- Department of Endocrinology M, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No